CLINICAL TRIAL: NCT05530525
Title: Psychometric Evaluation of Commonly Used Measures in Patients With Stroke Using Medical Record Review
Brief Title: Psychometric Evaluation of Commonly Used Measures in Stroke
Status: Completed | Type: Observational
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB110-263-B
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Test-retest reliability and responsiveness group (All of the data was collected from medical record): All the participants received conventional rehabilitation (e.g., occupational therapy, physical therapy, or speech therapy) or other interventions (e.g., acupuncture).
  Interventions: Diagnostic Test: The Computerized Adaptive Testing system of the Functional Assessment of Stroke; Diagnostic Test: The Barthel Index; Diagnostic Test: The National Institutes of Health Stroke Scale

INTERVENTIONS:
Diagnostic Test: The Computerized Adaptive Testing system of the Functional Assessment of Stroke — The Computerized Adaptive Testing system of the Functional Assessment of Stroke comprises 58 items. The items were selected from four well-known physical function measures for patients with stroke: 26 items from the Fugl-Meyer Assessment-Upper limb, 11 items from the Fugl-Meyer Assessment-Lower limb, 12 items from the Postural Assessment Scale for Stroke Patients, and 9 items from the Barthel Index. These items evaluate motor control, postural control, and activity of daily living functions in patients with stroke. Results are automatically reported as Rasch scores (i.e., the minimum and maximum values are negative and positive infinity, respectively). A higher score indicates greater physical functions.
Diagnostic Test: The Barthel Index — The Barthel Index has 10 items, and the total score ranges from 0 to 100. Higher score indicates less disability on activity of daily living functions.
Diagnostic Test: The National Institutes of Health Stroke Scale — The National Institutes of Health Stroke Scale comprises 11 items and was used to monitor the severity in the patients with stroke. The total score ranges from 0 to 42, with a higher score indicating greater severity. A National Institutes of Health Stroke Scale score of 1-5 indicates mild severity; 6-14, mild to moderate severity; 15-24, severe severity; and equal to or greater than 25, very severe severity.

SUMMARY:
Purposes: The aim of this study is to examine the psychometric properties (e.g. test-retest reliability, random measurement error, practice effect, and responsiveness) of the commonly used measures in patients with stroke using medical record review.

The investigators anticipate reviewing 1000 stroke patients' medical record from a medical center in Taiwan. The medical record will be reviewed by an experienced and well-trained occupational therapist.

DETAILED DESCRIPTION:
The investigators anticipate reviewing 1000 stroke patients' medical record (from 2018/6/1 to 2021/6/30) from a medical center in Taiwan. The medical record will be reviewed by an experienced and well-trained occupational therapist. The study was approved by the local institutional review board. Because the targeted populations for examining the test-retest reliability and responsiveness were different, the inclusion criteria were listed separately below.

Test-retest reliability Chronic stroke patients' data was reviewed to examine the test-retest reliability. The participants met the following criteria: (1) diagnosis of cerebral hemorrhage or cerebral infarction, (2) age ≥ 20 years, and (3) stroke onset ≥ 6 months (first and recurrent stroke included).

Responsiveness Subacute stroke patients' data was reviewed to examine the responsiveness. The participants met the following criteria: (1) diagnosis of cerebral hemorrhage or cerebral infarction, (2) age ≥ 20 years, and (3) stroke onset < 3 months (first and recurrent stroke included).

ELIGIBILITY:
Inclusion criteria for test-retest reliability group (Chronic stroke patients' medical record was reviewed to examine the test-retest reliability) :

* Cerebral hemorrhage or cerebral infarction.
* Age ≥ 20 years.
* Stroke onset ≥ 6 months (first and recurrent stroke included).

Inclusion criteria for responsiveness group (Subacute stroke patients' medical record was reviewed to examine the responsiveness):

* Cerebral hemorrhage or cerebral infarction.
* Age ≥ 20 years.
* Stroke onset < 3 months (first and recurrent stroke included).

Exclusion criteria

• Patients' diagnosis is not stroke.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the data was from the medical record (from 2018/6/1 to 2021/6/30) from the Department of Physical Medicine and Rehabilitation at a medical center in Taiwan.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The computerized adaptive testing system of the functional assessment of stroke | The repeated assessments were performed at an one-month interval.
  The Computerized Adaptive Testing system of the Functional Assessment of Stroke comprises 58 items. The items were selected from four well-known physical function measures for patients with stroke: 26 items from the Fugl-Meyer Assessment-Upper limb, 11 items from the Fugl-Meyer Assessment-Lower limb, 12 items from the Postural Assessment Scale for Stroke Patients, and 9 items from the Barthel Index. These items evaluate motor control, postural control, and activity of daily living functions in patients with stroke. Results are automatically reported as Rasch scores (i.e., the minimum and maximum values are negative and positive infinity, respectively). A higher score indicates greater physical functions.
The Barthel Index | The repeated assessments were performed at an one-month interval.
  The Barthel Index has 10 items, and the total score ranges from 0 to 100. Higher score indicates less disability on activity of daily living functions.
The National Institutes of Health Stroke Scale | The repeated assessments were performed at an one-month interval.
  The National Institutes of Health Stroke Scale comprises 11 items and was used to monitor the severity in the patients with stroke. The total score ranges from 0 to 42, with a higher score indicating greater severity. A National Institutes of Health Stroke Scale score of 1-5 indicates mild severity; 6-14, mild to moderate severity; 15-24, severe severity; and equal to or greater than 25, very severe severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Hualien County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided